CLINICAL TRIAL: NCT05220670
Title: Sarcopenia, Active Aging and Oral Microbiota in Older Adults. Effects of a High Intensity Exercises Program by Intervals
Brief Title: Sarcopenia, Active Aging and Oral Microbiota. Effects of HIIT in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University_Jaen
Record Dates: First submitted 2021-12-16; First posted 2022-02-02 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HIIT Group (Experimental): This group receives a training in which intervals of intense work and periods of active rest are combined using a cycle ergometer with an intensity of 85-95% of the maximum heart rate [MHR], followed by intervals of active rest of 3 minutes duration. at 50-70% MCF.
  Interventions: Other: HIIT
- MICT Group (Experimental): The participants will perform a training on the cycle ergometer with an intensity close to 70% FCM maintained for 40 minutes and will be controlled individually.
  Interventions: Other: MICT
- Control Group (No Intervention): The participants will receive advice on the general positive effects of the regular practice of physical activity, and will be given the guide of recommendations for the promotion of physical activity.

INTERVENTIONS:
Other: HIIT — It will be carried out after a 10-minute warm-up period with joint mobility exercises and dynamic stretching. The intervention will consist of a training in which intense work intervals and active rest periods are combined using a cycle ergometer. The session will be divided into 4 intervals of 4 minutes duration at an intensity of 85-95% of the maximum heart rate [MHR], individually controlled during all sessions (Polar Team pro®), followed by active rest intervals of 3 minutes duration at 50-70% FCM. After training, a 10-minute cool-down of gentle pedaling and joint range exercises will be carried out.
  Arms: HIIT Group
Other: MICT — Heating phase identical to the previous one. Subsequently, the participants will perform training on the cycle ergometer with an intensity close to 70% FCM maintained for 40 minutes and will be individually controlled (Polar Team pro®). The session will conclude with a cool-down phase identical to the previous one.
  Arms: MICT Group

SUMMARY:
To analyze the effects of a high intensity exercises program by intervals on sarcopenia, active aging and oral microbiota in older adults.

DETAILED DESCRIPTION:
All participants will be advised to lead healthy lifestyle habits according to the recommendations of the "Plan for the Promotion of Physical Activity and Balanced Eating of the Junta de Andalucía" http://www.juntadeandalucia.es/educacion/webporta/ishareservlet/content/86cf9950-abaa-403b-9fc3 9bc5ecae4614. A submaximal stress test will be performed at the beginning and end of the intervention. Before the test, the participants will become familiar with the measuring instrument with a warm-up that allowed them a gain in understanding the gear system. The test will start with a pedaling cadence of 50 revolutions, with an output power of 0 W, increasing by 25 W every 2 minute period. During the test there will be a continuous recording of blood pressure, heart rate and maximum oxygen consumption (VO2max). With this stress test, the aerobic and anaerobic threshold of each participant will be determined to mark the intensity of work at which each subject must perform physical activity in the intervention period.

The interventions of the 2 experimental groups are carried out with a frequency of 3 weekly trainings, for a total period of 16 weeks. The intensity of the training will be assigned to each subject individually based on the stress test performed in the previous phase. Experimental group 1 (HIIT): The HIIT protocol will be carried out after a 10-minute warm-up period with joint mobility exercises and dynamic stretching. The intervention will consist of training in which intense work intervals and active rest periods are combined using a cycle ergometer. The session will be divided into 4 intervals of 4 minutes duration at an intensity of 85-95% of the maximum heart rate [HRM], individually controlled during all sessions (Polar Team pro®), followed by active rest intervals 3 minute duration at 50-70% FCM. After the training, there will be a 10-minute cool down of gentle pedaling and joint range exercises. Experimental group 2 (MICT): Heating phase identical to the previous one. Subsequently, the participants will perform a training on the cycle ergometer with an intensity close to 70% FCM maintained for 40 minutes and will be controlled individually (Polar Team pro®). The session will conclude with a cool down phase identical to the previous one. Control group (CTRL): The participants will receive general advice on the positive effects of the regular practice of physical activity, and they will be given the guide of recommendations for the promotion of physical activity published by the Junta de Andalucía: http: // www.juntadeandalucia.es/salud/servicios/contenidos/andaluciaessalud/docs/130/Guia_Recomendaciones_AF.pdf

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* SARC-F ≥4 or handgrip strength <16 kg for women and < 27 kg for men.
* Not being afflicted by any condition preventing physical activity.
* Not being engaged in regular physical activity >20 minutes and >3 days/week.
* Being able to communicate without difficulty.
* Being able to read and understand the informed consent form as well as the goals of the study.

Exclusion Criteria:

* Acute or terminal illness.
* Unstable cardiovascular conditions.
* Conditions or medical treatments affecting the normal production of saliva (i.e. autoimmune disorders such as Sjögren's syndrome or medications like anxiolytics or antidepressants).
* Being or having been medicated with antibiotics up to one month prior to the taking of samples.
* Alcohol abuse or regular drug abuse.
* Severe visual or auditory impairment.
* Being involved in a different research group with the potential to interfere in our results.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Handgrip Strength | Up to twelve weeks
  Dynamometer will be employed to assess handgrip Strength
Relative abundance | Up to twelve weeks
  Determination of the % of specific bacteria in each of the taxonomic levels (phylum, family, genus and species).
Biodiversity | Up to twelve weeks
  Alpha and beta diversity, have a great effect on our health, since greater microbiota diversity is related with health.
ABC-16 (Activities Specific Balance Confidence Scale) | Up to twelve weeks
  Questionnaire that assesses balance confidence in performing activities of daily living. It is calculated by adding up the 16 responses of the questionnaire, with 0 being the minimum score and 100 being the maximum score. The higher value represents a better result.
FES-I (Falls Efficacy Scale-International) | Up to twelve weeks
  Questionnaire that evaluates the fear of falling. The score ranges from 7 to 28 points. Higher values indicate more concern related to falls.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid evaluation of both the quality of sleep and the alterations that may affect it.
  It consists of a total of 19 questions, grouped into 10 questions. The 19 questions are combined to form seven domains (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use, and daytime dysfunction, adding up to a total score) with their corresponding score, each one of which shows a range between 0 and 3 points. The higher value represents a worse result. The higher value represents a worse result. Higher bases indicate poorer sleep.
HADS (The Hospital Anxiety And Depression) | Up to twelve weeks
  A reliable, valid and practical screening tool for identifying and quantifying anxiety and/or depression in non-patients. The test contains 14 items with a score from 0 to 3, of which 7 items refer to depression and 7 to anxiety. The total score is 0-21, where a higher score corresponds to worse symptoms of anxiety and depression.
Percent of Body Fat (%) | Up to twelve weeks
  Indicates the percentage of body fat to body weight.

SECONDARY OUTCOMES:
BMI (Body Mass Index) | Up to twelve weeks
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat.
TUG (Timed Up and Go test) | Up to twelve weeks
  Is a simple test used to assess a person's mobility and physical function.
Short Physical Performance Battery (SPPB) | Up to twelve weeks
  It is an instrument that evaluates three aspects of mobility: balance, gait speed and strength of the lower limbs or limbs to get up from a chair.
Stabilometric Platform | Up to twelve weeks
  instrument composed of resistive pressure sensors, used to measure the static or postural balance. The test was performed under both eyes-open and eyes-closed conditions.
FSS (Fatigue Severity Scale) | Up to twelve weeks
  A self-report scale describing the severity of fatigue and the impact of fatigue on activities of daily living. The test is made up of 9 items with 7 response possibilities, so that 1 and 7 correspond to the minimum and maximum severity respectively. The total score corresponds to the sum of all the items with a total score range that goes from 9 to 63.
SF-36 (The Short Form-36 Health Survey) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The test consists of 36 items that detect both positive and negative health states. The total score ranges from 0 to 100, where 0 represents the worst quality of life and 100 the best.
Percent of Body Fat (%) | Up to twelve weeks
  Indicates the percentage of body fat to body weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Andina Area University Foundation, Pereira, Colombia, Spain

REFERENCES:
- [Derived] Lavilla-Lerma ML, Aibar-Almazan A, Martinez-Amat A, Jimenez-Garcia JD, Hita-Contreras F. Moderate-intensity continuous training and high-intensity interval training modulate the composition of the oral microbiota of elderly adults: Randomized controlled trial. Maturitas. 2024 Jul;185:107973. doi: 10.1016/j.maturitas.2024.107973. Epub 2024 Mar 26. PMID 38579579